CLINICAL TRIAL: NCT03269513
Title: OBESITY IN SCHOOLCHILDREN OF BASIC EDUCATION: a Study Interdisciplinary Intervention - Phase III
Brief Title: OBESITY IN SCHOOLCHILDREN OF BASIC EDUCATION - Phase III 2017
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Santa Cruz do Sul (Other)
Responsible Party: Principal Investigator, Miria Suzana Burgos, Principal Investigator, University of Santa Cruz do Sul
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UNISC
Record Dates: First submitted 2017-08-18; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Obesity; Overweight; Adolescent Obesity; Exercise
MeSH Terms: conditions — Obesity; Overweight; Pediatric Obesity; Motor Activity | interventions — Exercise; Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Adolescent Obesity
  The exercise program, nutritional counseling and oral health will last for five to three months and will be held in the gym and rooms of the University of Santa Cruz do Sul (UNISC).
  The sessions will last two hours (one hour of physical exercise and the second time divided into nutritional counseling, postural, psychological and oral) with a frequency of three times a week.
  Interventions: Behavioral: Physical Exercise
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Physical Exercise — The sessions will last two hours (one hour of physical exercise and the second time divided into nutritional counseling, postural, psychological and oral) with a frequency of three times a week.
  Other Names: Nutritional counseling; Psychological counseling
  Arms: Intervention group

SUMMARY:
The study aims to evaluate the possible effects of an exercise program, nutritional and psychological, postural orientation and guidance of oral health on body composition, physical activity levels and lifestyle, physical fitness and health and motor performance, the factors risk of cardiovascular disease, eating habits, the cognition levels, the psychological profile, the body posture of children and adolescent with overweight and obesity, considering the presence of risk genotype associated with the development of obesity. In addition, identify the effects of orientation for oral health on the quality of life and healthy oral habits.

ELIGIBILITY:
Inclusion Criteria:

* The official signing the informed consent and informed;
* The student with 12 years or older must sign the consent term;
* Age range: 10 to 17;
* Gender: male and female;
* No contraindications for blood collection;
* No distinction in relation to social class, ethnicity or color;
* To have a BMI greater than 85th percentile;
* Do not be participating in any other exercise program and dietary intervention;
* Participate in the clarification meetings on the project, when the head of the student is committed to the project, the following: a) assume responsibility for bringing to the UNISC (building 42) and refer to their home, the participant student of this study, both in the days of assessment (testing and completion of the data collection instruments), as in the days of intervention: 2nd, 4th and 6th fairs, from 14h to 16h, including 15 minutes in advance to the host, call and guidance students;
* Participate in intervention sessions during the period of 2 hours daily, the established days, following the guidelines given by the coordination of the project and the professionals of Physical Education, Nutrition, Psychology, Pharmacy, Physiotherapy, Medicine, Nursing and / or another area of health / education that can contribute to achieving the objectives of the intervention project;
* Participate in the assessments and reassessments as protocols established by the project.

Exclusion Criteria:

* Students who submit a frequency less than 70% stake in the intervention;
* Students who present contraindication to the practice of physical activity during the program implementation period;
* Students who choose not to continue with the treatment of intervention proposed by the program;
* Be in possession of any kind of illness, abnormality or health problem such as:

  * Hypertension untreated, Kidney diseases, Cardiac disorders, chronic renal failure, genetic diseases that have congenital malformations and mental retardation as Turner syndrome, Klinefelter syndrome and Down syndrome or cognitive impairment. And do not be carrying transmitted diseases vertically (from mother to child) with anatomical deformations caused by the interference of the pathogenic agent in the development process, as Congenital Toxoplasmosis (hydrocephalus, cerebral calcification, mental retardation, acute myocarditis, retinochoroiditis, strabismus, microphthalmia ), Rubella Syndrome, congenital (deafness, congenital cataracts, heart defects, microcephaly and mental retardation) congenital Syphilis (bone deformities, keratitis, deafness and mental retardation), cytomegalovirus infection congenital (microcephaly, intracranial calcifications and sensorineural deafness), because these subjects they need special care medical and/or service people trained for the specific purposes.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2017-11-23 (Estimated); Study Completion 2017-12-08 (Estimated)

PRIMARY OUTCOMES:
Change from body mass index (BMI) at 3 months | Baseline and 3 months.
  Weight and height will be evaluated early in the morning in a fasting state, with the student wearing light clothing and shoes. The BMI will be classified as normal BMI, overweight or obesity.The BMI will be classified according to the percentage curves of the Centers for Disease Control and Prevention / National Center for Health Statistics (CDC/NCHS) (2010) according to gender and age, considering the low weight (<p5), normal weight (p5 and <p85), overweight (p 85 and <p 95) and obesity (p 95).

SECONDARY OUTCOMES:
Change from the percentage of body fat at 3 months | Baseline and 3 months.
  To measure body fat percentage (BF%), a Lange (Beta Technology Incorporated) compass will be used to measure triceps and subscapular skinfolds. The equation of Slaughter et al. (1998) will be applied, and data will be classified according to Lonman's data, as mentioned by Heyward and Stolarczyk (2000).
Change from the waist circumference (WC) at 3 months | Baseline and 3 months.
  Waist circumference (WC) was measured with an inelastic tape, using the narrowest part of the trunk between the ribs and the iliac crest and the hip at the greater trochanter level as references. The subjects were then classified according to Taylor et al. (2000), defining the normal circumference percentile as <80 and obesity percentile as >80 according to gender and age.

CONTACTS AND LOCATIONS:
Overall Officials: Miria S Burgos, Dra, Principal Investigator — Universidade de Santa Cruz do Sul
Locations (1):
- Universidade de Santa Cruz do Sul, Santa Cruz do Sul, Rio Grande do Sul, Brazil